CLINICAL TRIAL: NCT02463669
Title: The Use of Point-of-Care Ultrasound in the Diagnosis of Acute Infectious Mononucleosis in the Emergency Department
Status: Terminated | Type: Observational
Why Stopped: COVID pandemic
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Laurie Robichaud, Laurie Robichaud, MD, Jewish General Hospital
Other Study IDs: POCUSIM01
Record Dates: First submitted 2015-05-31; First posted 2015-06-04 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Infectious Mononucleosis; Splenomegaly
Keywords: Point-of-care ultrasound
MeSH Terms: conditions — Infectious Mononucleosis; Splenomegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Point-of-care ultrasound — Enrolled patients will undergo POCUS of the spleen by the treating emergency physician (resident, fellow or attending). Canadian Emergency Ultrasound Society (CEUS) certified residents, fellows and attending physicians will conduct the bedside ultrasonography after receiving specific training for the purposes of this study. The spleen will be assessed using a curved 2-6 Megahertz (MHz) transducer with the participant in the supine position. The cranio-caudal splenic length will be measured and its maximum dimension will be recorded on the standardized study data sheet.

SUMMARY:
The purpose of this study is to determine if splenomegaly on point-of-care ultrasound (POCUS) is an accurate and user-friendly surrogate to the heterophile antibody test and Epstein-Barr Virus (EBV) serologies to diagnose acute mononucleosis infection in patients presenting with sore throat to the Emergency Department (ED).

DETAILED DESCRIPTION:
The investigators seek to determine whether the presence of splenomegaly on POCUS can accurately diagnose acute infectious mononucleosis in symptomatic ED patients, and determine the feasibility of performing point-of-care ultrasound for splenomegaly by emergency physicians in the emergency department setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 10 and 35 year-old presenting to the ED with suspected acute infectious mononucleosis

Exclusion Criteria:

* Chronic infectious disorders (eg. tuberculosis, malaria, HIV, syphilis)
* Inflammatory disorders (eg. sarcoidosis, amyloidosis, systemic lupus erythematosus, Felty syndrome)
* Proliferative disorders (eg. lymphoma, leukemia, essential thrombocytopenia, polycythemia vera)
* Congestive disorders (eg: cirrhosis, portal hypertension, right heart failure, congenital heart disease)
* Chronic haemolytic anemia (eg. sickle cell, thalassemia, hereditary spherocytosis)
* Storage diseases (eg. Gaucher, Niemann-Pick)
* Splenectomy
* Inability to give informed consent

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Convenience sample of patients between July 2016 and October 2017. Inclusion criteria are patients aged between 10 and 35 year-old presenting to the ED with suspected acute infectious mononucleosis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-04; Primary Completion 2020-10-04 (Actual); Study Completion 2020-10-04 (Actual)

PRIMARY OUTCOMES:
Presence of splenomegaly (maximal splenic cranio-caudal length) on point-of-care ultrasound | 12 months
  Splenomegaly is defined as a splenic length of > 11.5 centimetres (cm) for 10-12 year-old patients, > 12 cm for 12-15 year-old patients, > 12 cm for 15-35 year-old female patients, and > 13 cm for 15-35 year-old male patients.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - CHU Sainte-Justine, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided